CLINICAL TRIAL: NCT03752983
Title: Chemokine CXCL13 as a Marker of Disease Activity in Systemic Lupus Erythematosus
Brief Title: Chemokine (CXCL13) as Anew Marker in Diagnosis of SLE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Khamis Mohamed, Assuit lecturer, Assiut University
Other Study IDs: CXCL13 in SLE
Record Dates: First submitted 2018-11-22; First posted 2018-11-26 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-11

CONDITIONS: Systemic Lupus
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: patients with SLE
  Interventions: Diagnostic Test: blood samples
- controls: Healthy people
  Interventions: Diagnostic Test: blood samples

INTERVENTIONS:
Diagnostic Test: blood samples — blood samples

SUMMARY:
Systemic lupus erythematosus (SLE) is systemic autoimmune disease characterized by various immunological abnormalities, including dysregulated activation of both T and B lymphocytes with overt production of autoreactive antibodies.The chemokine CXC ligand 13 protein (CXCL13), also known as B cell-attracting chemokine-1 (BAC-1) or B lymphocyte chemoattractant (BLC), CXCL13 serum levels were correlated with disease activity using the SLE Disease Activity Index (SLEDAI) and to lupus nephritis

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is systemic autoimmune disease characterized by various immunological abnormalities, including dysregulated activation of both T and B lymphocytes with overt production of autoreactive antibodies . Lupus nephritis (LN) is the most common and serious complication in SLE patients characterized by proteinuria, hematuria, drop glomerular filtration rate, or renal dysfunction . It is known that B lymphocytes are involved in the pathogenesis of systemic lupus erythematosus in autoantibody-dependent mechanisms . The chemokine CXC ligand 13 protein (CXCL13), also known as B cell-attracting chemokine-1 (BAC-1) or B lymphocyte chemoattractant (BLC), is a CXC subtype member of the chemokine superfamily. The receptor of CXCL13 is CXCR5, which is normally expressed on mature B cells and follicular T helper cells (Tfh). It has been demonstrated that CXCL13 is sufficient to induce secondary lymphoid tissues in peripheral organs. It is well known that different chemokines are involved in the pathogenesis of LN by orchestrating proinflammatory microenvironments, recruiting immune cell subsets into the kidney and by inducing local activation of immune effector cells . Local B-cell infiltration and related abnormal expression of ectopic lymphoid tissue (ELT) in the renal tissues of LN mice models was related to the severity of renal impairment .

Of interest, in regions of B cell infiltration a higher expression level of CXCL13 was found. Most B cells in this region expressed the corresponding receptor CXCR5, also supporting the hypothesis that CXCL13 induces B cell infiltration into the kidneys via its receptor CXCR5 .

In one study on 91Caucasian patients, CXCL13 serum levels were correlated with disease activity using the SLE Disease Activity Index (SLEDAI) and to lupus nephritis. It was found that serum CXCL13 levels correlated well with SLEDAI and median CXCL13 concentrations were higher in patients with renal involvement .

ELIGIBILITY:
Inclusion Criteria:

* SLE patients diagnosed according to ACR

Exclusion Criteria:

* patient with other autoimmune diseases.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: two groups: 46 patients with SLE 40 healthy people
Sampling Method: Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
to measure the level of cxcl13 in SLE | Baseline
  to differentiate the level of (cxcl13) between healthy individuals and patients with SLE

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmadpoor P, Dalili N, Rostami M. An update on pathogenesis of systemic lupus erythematosus. Iran J Kidney Dis. 2014 May;8(3):171-84. PMID 24878938